CLINICAL TRIAL: NCT01377298
Title: A Phase II Study of Pazopanib in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Refractory to Platinum-Based Chemotherapy
Brief Title: Pazopanib in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Ruey-Long Hong, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201007042M
Record Dates: First submitted 2011-05-16; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib (Experimental): Single arm study, pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — 200mg/tablet, 800mg/day PO.

SUMMARY:
Because of the advantageous activity against VEGF-C and FGF pathways and favorable toxicity profile comparing with sunitinib, the investigators plan this phase II trial of pazopanib in cisplatin-refractory recurrent or metastatic HNSCC.

DETAILED DESCRIPTION:
Pazopanib, a tyrosine kinase inhibitor targets VEGFR1/2/3, PDGFR alpha & beta, c-KIT, and FGFR1/3 to inhibit angiogenesis. The phase II trial in advanced RCC (previous cytokine therapy in 25 % of patients) yielded good clinical benefits (response rate 34.6%; disease control 79.8%) with durable activity (progression-free to near 1 year) and acceptable toxicity. The randomized phase III trial in advanced RCC are ongoing and interim analysis revealed prolonged progression-free survival in pazopanib group compared with placebo group. Pazopanib is an active multi-targeted tyrosine kinase inhibitor needed to broaden it new indications to treat cancers. VEGF-C and FGF pathways are also important in the angiogenesis, metastasis, invasion, and cancer stem cell renewal in HNSCC. Pazopanib can also inhibit these two pathways and might offer much more suppression on tumor angiogenesis and growth in HNSCC compared with sunitinib. Common side effects of pazopanib are grade I to II diarrhea, hypertension, hair color change, and nausea, which are all manageable. Because of the advantageous activity against VEGF-C and FGF pathways and favorable toxicity profile comparing with sunitinib, we plan this phase II trial of pazopanib in cisplatin-refractory recurrent or metastatic HNSCC.

Serum inflammation markers, like IL-6 (esp. in inflammation- mediated cancers, like virus- related hepatocellular carcinoma and HNSCC), and host/tumor VEGF/VEGFR2 polymorphism attracted much attention in tumor angiogenesis dependence and response prediction of anti-angiogenesis treatments, in addition to previously described sVEGFR2 and circulating endothelial progenitors(CEP) in the phase II trial of RCC. We will study serum IL-6/VEGF/sVEGFR2/CEP and host/tumor VEGF/VEGFR2 polymorphism for prognosis and response correlation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed HNSCC.
2. Recurrent or metastatic setting, refractory to previous cisplatin or carboplatin-based chemotherapy.
3. At least one measurable lesion (according to RECIST v 1.1 criteria).
4. Eastern Cooperative Oncology Group performance status 0 to 2.
5. Age>18y/o,<=70y/o.
6. Adequate bone marrow, hepatic, and renal functions as evidenced by the following:

   * Absolute neutrophil count>=1,500 cells/L, platelet count>=100,000 cells/L, and hemoglobin>=9 g/dL.
   * Total bilirubin<=1.5 X ULN, AST/ALT<=3.0 X ULN
   * Creatinine<=1.5 mg/dL.
7. Informed consent, obtained in writing.

Exclusion Criteria:

1. Second malignancy.
2. Locoregional recurrence amenable to definite surgery or radiation again.
3. Brain/meningeal metastasis with IICP or bone metastasis with spinal cord compression.
4. Pregnancy or nursing women.
5. Having received more than two prior lines of intravenous chemotherapy in the palliative setting.
6. Having received antiangiogenesis agent in the palliative setting.
7. Having received chemotherapy or radiation therapy or surgery within 3 weeks.
8. Major systemic diseases those are inappropriate for systemic chemotherapy according to clinician's professional judgment.
9. Mental status not fit for clinical trials.
10. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

    * Active peptic ulcer disease
    * Known intraluminal metastatic lesion/s with risk of bleeding
    * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
    * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
11. Corrected QT interval (QTc)>480 msecs using Bazett's formula.
12. Poorly controlled hypertension defined as SBP>=140 mmHg or DBP>=90mmHg
13. Concomitant diseases that might be aggravated by investigational drugs:

    * Active or non-controlled infection.
    * Severe upper gastrointestinal bleeding.
    * History of any one or more of the following cardiovascular conditions within the past 12 months:
    * Cardiac angioplasty or stenting,
    * Myocardial infarction,
    * Unstable angina,
    * Symptomatic peripheral vascular disease,
    * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
14. Hemoptysis within 6 weeks of first dose of Pazopanib, prior major surgery within 4 weeks of first dose of Pazopanib, or presence of any non-healing wound/fracture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Evaluable for response: From the RECIST 1.1 paper,all patients included in the study must be accounted for in the results, even if there are major protocol treatment deviations or if they are not evaluable.

SECONDARY OUTCOMES:
disease control rate (CR+PR+SD), | 1 year
  Patients who receive at least 3 days of pazopanib will be included in the baseline, dosing and safety summaries. The primary calculation of complete response rate will be based on all response-evaluable patients.
Tumor Necrosis Ratio | 1 year
  Tumor Necrosis Ratio: On contrast enhanced T1WI, (CE-T1WI), manual delineation of the area of necrosis and entire tumor is performed on the central tumor-containing slice with the areas of necrotic center and entire tumor automatically generated. The tumor necrosis ratio is defined as the area of necrotic center over that of the entire tumor.
  (<25%, <50%, <75%, or >75%)
progression-free survival | 1 year
overall survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan